CLINICAL TRIAL: NCT02596880
Title: Sustained Viral Response Rate in 100 Subjects With Cirrhosis Due to Hepatitis C Treated With 12 Weeks of Sofosbuvir, Daclatasvir and Ribavirin
Brief Title: Sofosbuvir, Daclatasvir, Ribavirin for Hepatitis C Virus (HCV) Cirrhotics
Acronym: SD100
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Malekzadeh, MD, Professor of Gastroenterology and Hepatology, Tehran University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 94-02-159-30278
Record Dates: First submitted 2015-11-03; First posted 2015-11-04 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Hepatitis C; Cirrhosis
Keywords: Hepatitis C; Cirrhosis; Sofosbuvir; Daclatasvir; Ribavirin
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Sofosbuvir; daclatasvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Subjects will receive sofosbuvir, daclatasvir and ribavirin
  Interventions: Drug: Sofosbuvir; Drug: Daclatasvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Sofosbuvir — 400 mg, included in a combination pill (Sovodak) with 60 mg daclatasvir
  Other Names: Sovodak
Drug: Daclatasvir — 60 mg, included in a combination pill (Sovodak) with 400 mg sofosbuvir
  Other Names: Sovodak
Drug: Ribavirin — 1000 mg/day if <75 kg, 1200 mg/day for >75 kg. Divided into two daily doses
  Other Names: RBV

SUMMARY:
The investigators will treat 100 patients with cirrhosis due to hepatitis C with sofosbuvir 400 mg daily, daclatasvir 60 mg daily and weight-based ribavirin (1000 mg/d if <75 kg, 1200 mg/d if >75 kg, divided in two daily doses) for 12 weeks and calculate the sustained viral response rate at 12 weeks.

DETAILED DESCRIPTION:
Cirrhosis due to Hepatitis C presents a rather difficult treatment problem as many cannot tolerate interferon, the previous standard of treatment. The new direct acting antivirals have provided these patients with a new hope. One such combination is sofosbuvir (SOF) 400 mg and daclatasvir (DCV) 60 mg given once daily with or without weight-based ribavirin (RBV) for 12 or 24 weeks. The current recommendation for cirrhotics is SOF/DCV/RBV for 24 weeks but that recommendation is based on the lack of data for shorter periods. In order to evaluate the response rate to the combination of SOF/DCV/RBV the investigators decided to treat 100 HCV cirrhotics with this combination for 12 weeks. Subjects include genotype 1 and 3 patients, the prevalent genotypes in Iran. Patients with Model for End stage Liver Disease (MELD) > 20 are excluded. The investigators will calculate the sustained viral response rate at 12 weeks (SVR12).

ELIGIBILITY:
Inclusion Criteria:

* Positive qualitative HCV RNA test on two occasions at least 6 months apart
* Cirrhosis proven by either of: 1. Liver biopsy, 2. Liver elasticity > 12 kilopascal (KPa), 3. Clinical certainty (ascites, splenomegaly, small liver, low albumin, low platelet)

Exclusion Criteria:

* Renal failure (eGFR < 30 cc/min),
* MELD score > 20,
* Child's C (CTP score > 12),
* Heart rate < 50/min,
* Taking amiodarone

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
The sustained viral response rate | week 24 (12 weeks after end of treatment)
  Qualitative HCV RNA polymerase chain reaction (PCR)

SECONDARY OUTCOMES:
Adverse drug events | week 2, 4, 8, 12, 24
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Reza Malekzadeh, M.D., Study Chair — Tehran University of Medical Sciences
Locations (1):
- Shariati Hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No